CLINICAL TRIAL: NCT02802579
Title: ECG Triggered Dual Source CT for Non-invasive Pre-operative Cardiac Imaging in Morbid Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Sebastian Leschka, MD, Attending Physician, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RAD0701
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Obesity, Morbid
Keywords: obesity; dual source CT; coronary CT angiography; prognosis; bariatric surgery; gastric bypass surgery; coronary arterial disease; major adverse coronary event
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: standard protocol (Active Comparator): Standard dual-source computed tomography coronary angiography protocol
  Interventions: Radiation: standard protocol
- B: enhanced protocol (Experimental): enhanced dual-source computed tomography coronary angiography protocol
  Interventions: Radiation: enhanced protocol
- C: enhanced obesity protocol (Experimental): enhanced obesity-mode dual-source computed tomography coronary angiography protocol
  Interventions: Radiation: enhanced obesity protocol

INTERVENTIONS:
Radiation: standard protocol — tube voltage: 120 kV current time product: 350 mAs/rotation rotation: 90° (with two detectors in a 90° angle)
  Other Names: dual source computed tomography coronary angiography
  Arms: A: standard protocol
Radiation: enhanced protocol — tube voltage: 140 kV current time product: 350 mAs/rotation rotation: 90° (with two detectors in a 90° angle)
  Other Names: dual source computed tomography coronary angiography
  Arms: B: enhanced protocol
Radiation: enhanced obesity protocol — tube voltage: 140 kV current time product: 350 mAs/rotation rotation: 180° (with two detectors in a 90° angle)
  Other Names: dual source computed tomography coronary angiography
  Arms: C: enhanced obesity protocol

SUMMARY:
Coronary arterial disease is a risk factor for bariatric surgery and might be a predictor for later major adverse coronary events. Diagnosis of coronary arterial disease would thus be desirable for obese patients, however percutaneous angiography is an invasive procedure and associated with a certain morbidity in obese patients. In this study the investigators would like to assess whether dual source CT angiography can be used for diagnosis of coronary arterial disease in severely obese patients and which settings yield the best image quality.

DETAILED DESCRIPTION:
Obesity is a major health problem in many countries and a major risk factor for cardiovascular disease. Extreme obesity can be treated with surgery, however these procedures are associated with a certain surgery-related morbidity which increases with comorbidities, in particular coronary diseases. Thus, preoperative cardiac risk assessment would be desirable, however percutaneous coronary angiography is an invasive procedure with problems and complications in obese patients. A non-invasive alternative would be coronary dual-.source CT angiography (CCTA), however little experience exists in the application of CCTA in morbid obese patients. This study would like to address the following issues:

1. Comparison of image quality of coronary CT angiography using a dual source CT from obese patients using a special protocol (140 kV, 350 mAs) with images from historical controls from normal weight patients with a standard protocol (120 kV, 330 mAs).
2. Prediction of major adverse coronary events. Patients with a coronary stenosis in CCTA will be followed for any major adverse coronary events (details see Outcomes)
3. Is it possible to detect myocardial fat by a reduced CT density. Images from obese patients will be compared to historical controls from normal patients. Furthermore, is the myocardial CT density correlated with the BMI of obese patients?
4. Optimisation of scan protocol. Increasing the scanning angle beyond the standard 90° will reduce the signal noise at the cost of temporal resolution. Various scanning angles with be tested for an optimal combination of signal noise and temporal resolution.
5. Does the long QT-syndrome improve after bariatric surgery? It is assumed that the long QT-syndrome is a consequence of fattening of the myocardia. Is it possible to see a reduction of myocardial fattening and thus an improvement of the long QT-syndrome with CT during the follow-up after bariatric surgery?

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity (BMI >35 kg/m²)
* intention to undergo bariatric surgery
* increased risk for coronary artery disease (based on PROCAM score)

Exclusion Criteria:

* kidney insufficiency (serum creatinine >100 µmol/l, creatinine clearance <50 ml/min)
* allergy to iodine containing contrast agents
* hyperthyroidism
* metformin medication
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Image quality | 7 days
  Coronary arteries (with at least 1 mm diameter at their origin) were segmented according to the 15-segment model of the American Heart Association (Austen 1975). Subjective image quality was judged for each coronary artery segment on a 4-point scale (Leschka 2007) :
  1. = excellent;
  2. = good, minor artifacts;
  3. = fair, moderate artifacts but still diagnostic;
  4. = non-diagnostic
coronary artery stenosis | 7 days
  Significant coronary artery stenosis was defined as more than 50% narrowing of luminal diameter. Stenosis assessment was performed by a radiologist not involved in image quality assessment.

SECONDARY OUTCOMES:
Image noise | 7 days
  Image noise was determined as the standard deviation of the attenuation value in a region of 1 sq cm that was placed in the ascending aorta. The average of the attenuation in the left and right coronary artery were used for further calculations.
Signal-to-noise ratio (SNR) | 7 days
  SNR was determined by dividing mean attenuation by image noise
contrast-to-noise ratio (CNR) | 7 days
  Vessel contrast was calculated as the difference in the mean attenuation (in Hounsfield units) between the contrast-enhanced vessel lumen and the mean attenuation in the adjacent perivascular tissue. Attenuations were measured in a region in the proximal segment of the right coronary artery and in the left main artery, and were defined as large as possible, whereas avoiding calcifications and plaques. CNR was calculated as vessel contrast divided by image noise (Husmann 2006, Lembcke 2004).
Major adverse cardiovascular events (MACE) | 7 years
  Any of the following events:
  * death
  * non fatal myocardial infarction
  * late revascularization with percutaneous coronary intervention
  * coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Leschka, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austen WG, Edwards JE, Frye RL, Gensini GG, Gott VL, Griffith LS, McGoon DC, Murphy ML, Roe BB. A reporting system on patients evaluated for coronary artery disease. Report of the Ad Hoc Committee for Grading of Coronary Artery Disease, Council on Cardiovascular Surgery, American Heart Association. Circulation. 1975 Apr;51(4 Suppl):5-40. doi: 10.1161/01.cir.51.4.5. No abstract available. PMID 1116248
- [Background] Leschka S, Scheffel H, Desbiolles L, Plass A, Gaemperli O, Valenta I, Husmann L, Flohr TG, Genoni M, Marincek B, Kaufmann PA, Alkadhi H. Image quality and reconstruction intervals of dual-source CT coronary angiography: recommendations for ECG-pulsing windowing. Invest Radiol. 2007 Aug;42(8):543-9. doi: 10.1097/RLI.0b013e31803b93cf. PMID 17620936
- [Background] Husmann L, Alkadhi H, Boehm T, Leschka S, Schepis T, Koepfli P, Desbiolles L, Marincek B, Kaufmann PA, Wildermuth S. Influence of cardiac hemodynamic parameters on coronary artery opacification with 64-slice computed tomography. Eur Radiol. 2006 May;16(5):1111-6. doi: 10.1007/s00330-005-0110-4. Epub 2006 Jan 28. PMID 16607499
- [Background] Lembcke A, Wiese TH, Schnorr J, Wagner S, Mews J, Kroencke TJ, Enzweiler CN, Hamm B, Taupitz M. Image quality of noninvasive coronary angiography using multislice spiral computed tomography and electron-beam computed tomography: intraindividual comparison in an animal model. Invest Radiol. 2004 Jun;39(6):357-64. doi: 10.1097/01.rli.0000123316.10765.6c. PMID 15167102